CLINICAL TRIAL: NCT01852916
Title: Nasal High Frequency Oscillatory Ventilation (NHFOV) Versus Nasal Continuous Positive Airway Pressure (NCPAP) Ventilation: a Pilot Trial
Brief Title: NHFOV Versus NCPAP to Prevent Exubation Failure
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment rate
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Yaser Ali, Fellow, Neonatal-Perinatal Medicine, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2013: 040
Record Dates: First submitted 2013-04-17; First posted 2013-05-14 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: RDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal CPAP (Active Comparator): Nasal CPAP using Infant flow
  Interventions: Device: CPAP
- NHFOV (Experimental): Nasal High Frequency Oscillatory Ventilation using Dräger Babylog® VN500 ventilator machine
  Interventions: Device: NHFOV

INTERVENTIONS:
Device: CPAP — Nasal Continuous Positive Airway Pressure Ventilation using Infant Flow CPAP machine
  Arms: Nasal CPAP
Device: NHFOV — Nasal High Frequency Oscillatory Ventilation
  Arms: NHFOV

SUMMARY:
The purpose of the study is to assess whether nasal high frequency ventilation (NHFV) is superior to nasal continuous positive pressure (nCPAP) to prevent tracheal intubation and mechanical ventilation in preterm infants less than 28 weeks gestation following first attempt at extubation and removal from mechanical ventilation

DETAILED DESCRIPTION:
Extremely preterm infants frequently need to be placed back on invasive mechanical ventilation following initial attempts to remove them from this mode of respiratory support. Continued mechanical ventilation is thought to be the primary driver in the development of chronic lung disease and a major component in adverse developmental outcome of these infants. Infants fail their first trial of removal from ventilation because of apnea and respiratory failure. Animal studies and early clinical experience suggest that it is possible to effectively provide ventilation via high frequency nasal ventilation. In the animal models this mode of ventilation appears to provide for better lung development and less injury.

Nasal CPAP has been shown to improve the success rate of extubation from mechanical ventilation by preventing post extubation atelectasis with resultant improvements in gas exchange. However in many of the most premature infants, poorly developed control of respiratory drive is a major problem and despite treatment with caffeine, mechanical ventilation is needed. High frequency nasal ventilation may support ventilation enough during apneic periods to mitigate the need for traditional mechanical ventilation. Use of non-invasive modes may result in a decrease in the incidence and or severity of chronic lung problems and developmental disability of this group of infants.

Extremely premature infants (GA <28 weeks) less than 7 days old will be randomized to either NHFV or nCPAP following the first attempt at extubation and removal from mechanical ventilation. All infants will have received at least a loading dose of caffeine citrate (10 mg/kg of caffeine base equivalent prior to extubation. Initial nCPAP level will be determined by clinical staff but will be at least equal to the level of positive end expiratory pressure (PEEP) used during mechanical ventilation. A similar level of pressure will be used as initial mean airway pressure (MAP) in infants receiving HFNV.

The primary outcome will be need for reintubation during the first 7 days after extubation attempt due to preset criteria. Crossover to the other modality will not be allowed during this period. Infants may remain on HFNF beyond the 7 day primary endpoint if deemed necessary by the clinical staff. Weaning of HFNV to nCPAP will be allowed during the 7 day primary study period and reinstitution of HFNF will be allowed for those initially randomized to that mode of respiratory support.

The magnitude of the effect size cannot be determined as there are no studies to base a sample size calculation on. A pragmatic sample size of 20 infants was selected (10 in each arm) to allow estimation of any potential effect size. Further study(ies) will need to be performed to show conclusively efficacy (or lack) of NHFV to prevent post-extubation respiratory failure or its use in preventing chronic lung disease or improving developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newborn less than 28 weeks gestation at birth
* Intubated and ventilated in the first 24 hours of life
* Extubated in the first week of life
* Parental consent

Exclusion Criteria:

* Lack of parental consent
* Major congenital malformation
* Severe perinatal asphyxia
* Airway abnormalities
* Pneumothorax

Ages: 15 Minutes to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | within 7 days post-extubation
  Newborns in both groups will be re-intubated within the study period if they have respiratory failure defined as arterial or capillary gas with pH < 7.20 or PCO2 > 60, oxygen requirement ≥ 35%, or recurrent or severe apnea (12 documented apneas within 24 hours or single apnea requiring positive pressure ventilation).

SECONDARY OUTCOMES:
Changes in capillary pCO2 after extubation | Within 7 days post-extubation
  capillary pCO2 values will be measured after extubation. Timing and frequency of blood gas sampling will be determined by clinical staff caring for infant and will not be specified by study protocol.
pneumothorax | duration of use of positive pressure or reintubation which ever is shorter
  incidence of pneumothorax during use of either nasal CPAP or high frequency nasal ventilation will be documented.
intraventricular hemorrage (IVH) | first 2 weeks of life
  Infants will be screened for IVH per routine clinical care. Incidence of total IVH and severe IVH will be compared between treatments.
feeding tolerance | 3 weeks
  The time to achieve full enteral feeding (135 ml/kg/d) will be compared for both treatments

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Baier, M.D., Study Director — HSC Neonatology
Locations (2):
- Canada (2):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Center, NICU, Winnipeg, Manitoba